CLINICAL TRIAL: NCT00913471
Title: Biomarkers for Pain in Spinal Cord Injury (SCI) Patients
Acronym: SCI Pain
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The Institute for Rehabilitaion and Research Foundation (Other)
Responsible Party: Principal Investigator, Georgene Hergenroeder, Associate Professor, Neurosurgery, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-MS-07-0452
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Spinal Cord Injury; Neuropathic Pain
Keywords: Spinal cord injury; SCI; Neuropathic pain; Pain
MeSH Terms: conditions — Neuralgia; Spinal Cord Injuries; Pain | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples (120 subjects) and skin tissue biopsy (20 subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Acute-Longitudinal SCI
  Interventions: Other: blood samples
- Chronic SCI
  Interventions: Other: blood samples
- Healthy volunteers
  Interventions: Other: blood samples

INTERVENTIONS:
Other: blood samples — Chronic patients - a one time blood sample (12 mL) and questionnaire; 10 subjects will donate a 3-5mm skin tissue sample.
  Longitudinal Patients - 5 blood samples (12 mL each, totaling 60 mL at the following time points: within 48 hours, one week, one month, 6 months and 18 months post injury to coincide with standard visits) and questionnaire. 10 subjects will donate a 3-5mm skin sample.
  Healthy, pain free volunteers - a one time blood sample (12 mL), vital signs per standard CRU protocol and questionnaire confirming they are healthy.

SUMMARY:
The investigators propose to compare plasma protein profiles for SCI patients with/without chronic neuropathic pain in order identify biomarker(s) that are associated with this medical condition. Secondly, the investigators propose to identify a temporal relationship to initial SCI at which these biomarkers manifest.

Our working hypothesis is that sustained alterations in specific inflammatory molecules are associated with chronic neuropathic pain following SCI, and that their plasma levels can serve as biomarkers to identify patients at risk for the development of neuropathic pain.

Additionally the investigators are collecting skin tissue biopsy samples from patients following acute and chronic spinal cord injury to create vector-free human iPS cells from fibroblasts by direct delivery of reprogramming proteins.

ELIGIBILITY:
A. Chronic Patients

Inclusion:

1. Two or more years post traumatic SCI with deficit

Exclusion:

1. < 18 years of age
2. Evidence of brain injury on computed tomography (CT) (SCI patients need to be able to comply with completing the pain survey)
3. Other medical condition that accounts for chronic pain (i.e. diabetic neuropathy, renal insufficiency, multiple sclerosis, HIV associated neuropathy, alcohol-related neuropathy)
4. Temperature > 100.5°C
5. History of infection within the last 30 days (i.e. UTI, URI, pressure sore)
6. History of Pulmonary Embolus (PE) or deep vein thrombosis (DVT)
7. Inability to obtain informed consent
8. Psychiatric problems (patients need to be able to complete the pain survey)
9. Diagnosis or treatment of cancer in the last 5 years

B. Longitudinal, Prospective Cohort Patients:

Inclusion:

1. Initial traumatic SCI with deficit

Exclusion:

Same as listed above C. Healthy Volunteers Healthy volunteers include gender, age and race matched volunteers able to provide informed consent who have,

1. No significant medical history (pain free)
2. No recent infections
3. Take no medications
4. Fever free
5. Greater than 18 years old

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Acute and Chronic traumatic spinal cord injury patients and healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
To identify candidate biomarkers for pain in the chronic SCI samples. | two or more years post injury

SECONDARY OUTCOMES:
To identify the temporal relationship of the development of pain and the manifestation of the biomarkers identified | two or more years post injury

CONTACTS AND LOCATIONS:
Overall Officials: Georgene Hergenroeder, PhD, Principal Investigator — UTHSC-Houston
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.

REFERENCES:
- [Background] Hergenroeder GW, Moore AN, Schmitt KM, Redell JB, Dash PK. Identification of autoantibodies to glial fibrillary acidic protein in spinal cord injury patients. Neuroreport. 2016 Jan 20;27(2):90-3. doi: 10.1097/WNR.0000000000000502. PMID 26629661
- [Background] Hergenroeder GW, Redell JB, Choi HA, Schmitt L, Donovan W, Francisco GE, Schmitt K, Moore AN, Dash PK. Increased Levels of Circulating Glial Fibrillary Acidic Protein and Collapsin Response Mediator Protein-2 Autoantibodies in the Acute Stage of Spinal Cord Injury Predict the Subsequent Development of Neuropathic Pain. J Neurotrauma. 2018 Nov 1;35(21):2530-2539. doi: 10.1089/neu.2018.5675. Epub 2018 Jul 5. PMID 29774780